CLINICAL TRIAL: NCT06163144
Title: Risk Factors of Thrombocytopenia In Chronic Kidney Disease And Hemodialysis Patients In Assiut University Hospitals
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ata Kamel, resident doctor at internal medicine department, Assiut University
Other Study IDs: thrombocytopenia CKD
Record Dates: First submitted 2023-11-16; First posted 2023-12-08 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-11

CONDITIONS: Thrombocytopenia in CKD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients CKD 4, CKD 5 non- HD: chronic kidney disease patients non hemodialysis
  Interventions: Other: lab investigation
- Patients with ESRD on Regular -HD: end stage renal disease patients on hemodialysis
  Interventions: Other: lab investigation

INTERVENTIONS:
Other: lab investigation — Platlets count by : advia cell counter principles . This flow cytometry-based system uses light scatter, differential white blood cell (WBC) lysis, and myeloperoxidase and oxazine 750 staining to provide a complete blood cell count, a WBC differential, and a reticulocyte count. A cyanide-free method is used to measure hemoglobin colorimetrically.
  *Automated cell counters
  * Advia 2120 8 difference
  * PLT , parameters , MPV . Prothrombin time , prothrombin concentration , International normalized ratio , activated partial thromboplastin time . BUN, Serum Createnin Serum Albumin Serum Ca, Ph, PTH HBsAg, HCV - Abs Erythrocyte sedimintation rate ,C- reactive protein . 2.Specific lab: C3 - C4, Anti Neuclear Antibody, Anti douple stranded DNA , if suspect lupus . PCR for HCV or HBV serum lactate if sepsis is suspected. drugs level if Addiction is suspected.

SUMMARY:
factors contributing to thrombocytopenia in ESRD include uremia, blood loss, sepsis, and heparin treatment (2).

Haemodialysis (HD) has been also identified as a potential cause of thrombocytopenia due to the interaction of dialysis membranes with platelets, triggering adhesion, aggregation, and activation.

Renal replacement therapy has improved in recent decades, particularly with the use of synthetic and highly biocompatible dialyzer membranes. During hemodialysis treatment, patients are exposed to a variety of components of the dialysis circuit and thrombocytopenia is not uncommon

DETAILED DESCRIPTION:
Thrombocytopenia is defined as a platelet count below 150,000/mm3 and can result from decreased platelet production, increased platelet destruction, or splenic sequestration. The severity of thrombocytopenia is categorized as mild (platelet count above 70,000/mm3) or severe (platelet count below 20,000/mm3). While individuals with a count above 50,000/mm3 are often asymptomatic, severe cases can lead to various forms of bleeding, such as mucosal, intracranial, gastrointestinal, and genitourinary bleeding .

End-stage renal disease (ESRD) is associated with abnormalities in both platelet count and function. Etiological factors contributing to thrombocytopenia in ESRD include uremia, blood loss, sepsis, and heparin treatment .

Haemodialysis (HD) has been also identified as a potential cause of thrombocytopenia due to the interaction of dialysis membranes with platelets, triggering adhesion, aggregation, and activation.

Renal replacement therapy has improved in recent decades, particularly with the use of synthetic and highly biocompatible dialyzer membranes. During hemodialysis treatment, patients are exposed to a variety of components of the dialysis circuit and thrombocytopenia is not uncommon Platelets, derived from megakaryocytes, are cell fragments present in the bloodstream. After release from the bone marrow, they are stored in the spleen for 24 to 48 hours. The spleen holds around 30% of circulating platelets, which typically have a lifespan of about 7 days. Platelets are removed from the bloodstream by macrophages .Platelet count in normal conditions range from 150,000 to 450,000/mm in peripheral blood.

Decreased platelet count occurs due to Reduced bone marrow production, increased platelet destruction, and other factors like drugs or alcohol consumption contribute to decreased platelet count. An alteration in the number of megakaryocytes indicates changes in destruction or production . Hemodialysis can lead to a 15% reduction in platelet count during a session, with subsequent recovery after treatment due to factors such as adhesion and complement activation, regardless of the dialysis membrane material Heparin-induced thrombocytopenia (HIT) is a condition that results in a prothrombotic state, particularly impacting patients with chronic kidney disease (CKD) undergoing hemodialysis (HD).Heparin induced thrombocytopenia (HIT) occurs when antibodies to platelet factor 4 (PF4) and heparin complexes bind to the Fragment Crystalloid γRIIA receptors (FcγRIIA) on platelets and monocytes to begin a hypercoagulable state that may cause thrombosis. Antibodies to PF4-heparin complexes are frequently detected in patients treated with unfractionated heparin. Orthopedic surgery, lower platelet count and higher titer of PF4-heparin antibodies have been shown to be concurrent factors that increase the risk of thrombosis in HIT. Hemodialysis, autoimmune diseases, gout, heart failure, intravenous route of heparin and>5 days of heparin use were found to increase the risk of HIT diagnosis in medical patients . Substantial activation of platelets can occur in the course of hemodialysis. Platelet surface markers show evidence of platelet degranulation. Some activation occurs due to exposure of blood to the roller pump segment and microbubbles may play a rol Platelet activation seems to be reduced with reused dialyzers or with those containing synthetic versus cellulose membranes. Nevertheless, a substantial degree of platelet activation can be demonstrated with polysulfone and other synthetic membranes . the amount of activation may differ substantially among polysulfone membranes, depending on the manufacturer and the polyvinylpyrrolidone content. Platelet-platelet and platelet-leukocyte aggregates have been detected in the dialyzer blood outflow line and the consequences of these to the microcirculation are unknown. Typically, the platelet count decreases slightly during the first hour of dialysis, but mostly returns to initial values by the end of dialysis. Most recent cases of dialysis-associated thrombocytopenia have been with polysulfone membranes, especially polysulfone membranes sterilized by electron beam . Patients on HD also carry a greater risk of presenting with chronic hepatitis B virus (HBV) and hepatitis C virus (HCV) infection, with a much higher prevalence in developing countries . Thrombocytopenia is one of the most widespread complications of chronic viral hepatitis (CVH). It appears secondary to hypersplenism in cirrhosis, immune-mediated mechanisms, shear stress, hyperfibrinolysis, bacterial translocation, sepsis, viral suppression of platelet production in the bone marrow, and decreased thrombopoietin. Thrombocytopenia interferes with interferon during antiviral treatment . hemolytic uremic syndrome commonly presents with the triad of microangiopathic hemolytic anemia, thrombocytopenia, and renal function impairment without an antecedent hemorrhagic diarrhea. Less known are extrarenal complications due to abnormal vascular permeability, although these are a major cause of morbidity and mortality for the patients. Furthermore, it is increasingly recognized that the disease may present with hypertension or renal function impairment with no or mild thrombocytopenia and microangiopathic hemolytic anemia . Awareness of the full spectrum of atypical hemolytic uremic syndrome may facilitate its diagnosis and treatment before serious complications or death occurs . Sepsis is a global health burden that needs intensive medical care. Thrombocytopenia in sepsis is well known to increase morbidity as well as mortality. Several studies have been performed both in animal models and in humans to understand the mechanism by which sepsis causes thrombocytopenia . Recent studies have shown that inhibiting thrombocytopenia improves outcomes in sepsis patients. Understanding these mechanisms to identify targets in use of newer treatment modalities besides using resuscitation measures, antibiotics and removal of thrombocytopenia inducing agent could potentially help us improve outcomes in sepsis .

Drug-induced thrombocytopenia occurs when certain medicines destroy platelets or interfere with the body's ability to make enough of them. There are two types of drug-induced thrombocytopenia: immune and non-immune. If a medicine causes the body to produce antibodies, which seek and destroy the platelets, the condition is called drug-induced immune thrombocytopenia. Heparin, a blood thinner, is the most common cause of drug induced immune thrombocytopenia If a medicine prevents bone marrow from making enough platelets, the condition is called drug-induced nonimmune thrombocytopenia. Chemotherapy drugs and a seizure medicine called valproic acid may lead to this problem. Other medicines that cause drug-induced thrombocytopenia include: Furosemide, gold, NSAIDs, penicillin, quinidine,quinine ,Ranitidine ,sulfonamide ,Statins Platelet count is regularly low in patients after multiple trauma, mainly due to blood loss and dilution.

Thrombopoietin is the main regulator of the circulating platelet mass. Under several clinical conditions an inverse correlation between thrombocytopenia and the circulating platelet mass was reported. Since platelets bind and internalize thrombocytopenia, a platelet-dependent regulation of thrombocytopenia was suggested. Thus, acute blood loss should be accompanied by elevated thrombocytopenia Will be measured serum thrombocytopenia, platelets, interleukin-6 (IL-6) and vascular endothelial growth factor (VEGF) . In multiple traumatized patients low platelet count is followed by a rapid increase in serum TPO. This fits into the concept of a feedback regulation between circulating TPO and platelet mass.

ELIGIBILITY:
Inclusion Criteria:

* .Patient age between 18: 70 years old 2 .CBC with platelet count less than (80,000- 150,000) 3 .Hemodialysis duration > 6 months

Exclusion Criteria:

* .Decompensated liver disease. .known patients with idiopathic thrombocytopenia by bone marrow studies.

  * Known patients with multiple myeloma and blood malignancies ( leukaemia ,, lymphoma
  * Systemic lupus eryrthomatosis patients .Acute kidney injury patients .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Study population: 132 Patients divided into two groups Group A : including 54 Patients CKD 4, CKD 5 non- HD Group B : including 77Patients with ESRD on Regular -HD .
  According to CKD - staging by KDIGO 2012 / 2022:
  CKD 1 ≥ 90 ml / min ( normal or high ) CKD 2 :60 - 89 ml/min( mild decrease ) CKD 3a : 45 - 59 ml/min( mild to moderate decrease ) CKD 3b : 30 -44 ml/ min ( moderate to sever decrease ) CKD 4: 15 - 29 ml/min(sever decrease ) CKD 5 : < 15 ml/min( kidney failure ) .
Sampling Method: Non-Probability Sample
Enrollment: 132 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
platelets counts by manual ,direct ,and indirect | 1 year
  Manual Platelet counts Platelet counts can be done manually with a commercial diluting system, hemocytometer, and a microscope. These counts are less accurate than automated counts, because platelets can be difficult to distinguish from debris. Direct method Platelet count are done in the 5 intermediate square of the large central square using the HPO.Materials1. EDTA specimen of patient. Microscope. Reese and Ecker diluting fluid4. Hematocytometer5. RBC pipette with rubber tubing6. Cell counter Procedure. Indirect method PLATELET COUNT Compare to direct, it uses dilution of blood using RBC or WBC pipet and Neubauer Chamber Indirect, the platelets in RBC arecounted simultaneously in a bloodsmear, so there will be no dilution to lyseselectively the RBC and platlets .
albuminuria | 1 year
  A1 : < 30 mg / g or < 3 mg / mmol ( normal to mild increase ) A2 : 30 - 300 mg / g or 3-30 mg / mmol ( moderatly increase ) A3: > 300 mg / g or > 30 mg / mmol

SECONDARY OUTCOMES:
most frequent Risk factor of thrombocytopenia in chronic kidney diseases | 1 year
  as hemodialysis,

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah R, Haddad N, Vachharajani TJ, Asif A, Agarwal A. Thrombocytopenia in ESRD patients: epidemiology, mechanisms and interventional nephrology perspective. Semin Dial. 2014 Nov-Dec;27(6):618-25. doi: 10.1111/sdi.12199. Epub 2014 Feb 24. PMID 24612107
- [Background] Arepally GM. Heparin-induced thrombocytopenia. Blood. 2017 May 25;129(21):2864-2872. doi: 10.1182/blood-2016-11-709873. Epub 2017 Apr 17. PMID 28416511
- [Background] Arepally G, McKenzie SE, Jiang XM, Poncz M, Cines DB. Fc gamma RIIA H/R 131 polymorphism, subclass-specific IgG anti-heparin/platelet factor 4 antibodies and clinical course in patients with heparin-induced thrombocytopenia and thrombosis. Blood. 1997 Jan 15;89(2):370-5. PMID 9002937
- [Result] Gauer RL, Braun MM. Thrombocytopenia. Am Fam Physician. 2012 Mar 15;85(6):612-22. PMID 22534274